CLINICAL TRIAL: NCT06941090
Title: Nutrition, Gut Microbiota and Health : Feces Sample Collection in NutriNet-Santé Participants
Acronym: NUTRIGUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C21-60
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stool sampling (Experimental): The research consists in collecting stool samples from a sub-sample of participants already included in the NutriNet-Santé cohort. The stool collection will enable us to study the characteristics of the intestinal microbiota in relation to nutrition on the one hand, and health on the other, based on data collected during participation in the NutriNet-Santé cohort.
  Interventions: Other: sampling stool

INTERVENTIONS:
Other: sampling stool — Participants will receive a self-sampling stool kit with detailed instructions by mail to their home address. Samples will be mailed back by the participant to the treatment laboratory, which will determine the characteristics of their intestinal microbiota.

SUMMARY:
The gut microbiota is currently attracting increasing attention from the scientific community and also from the general public, as evidence of its role in human physiology has been highlighted. Microbial signatures have also been associated with various pathologies (e.g. obesity, diabetes, gastrointestinal disorders, neurodegenerative diseases), but the causality of these associations is still uncertain. Among the factors that may influence the composition of the gut microbiota (e.g. lifestyle, hygiene, medication, genetics, environment), nutrition would a major role. The major changes in lifestyle and diet observed over recent decades are strongly suspected of disrpting the host-gut microbiota balance.

In addition to their nutrient content, our diets also contain other bioactive compounds (e.g. polyphenols) and raise new issues (e.g. temporal structure of diets, food processing, presence of additives or contaminants such as pesticide residues, intake of dietary supplements, dietary exclusions, glycemic index) that is necessary to take into account. Thus, it is mandatory to explore and characterize in a more precise way, within large samples consisting of individuals with varied characteristics, the way in which the composition of the gut microbiota is influenced by the host's diet and its health consequences.

The aim of this research is therefore to study the links between nutrition, gut microbiota profiles and health. To do this, the research will implement large-scale stool sample collection from participants in the NutriNet-Santé cohort ("Nutrinautes"), thus constituting a "microbiota" sub-cohort.

A target of N=10,000 participants in the NutriNet-Santé cohort will be recruited on a voluntary basis. A selection will then be made among Nutrinautes willing to participate in the research (which may be more numerous than necessary) to maximize the diversity of profiles. Participants will be informed of their selection or non-selection by e-mail. A second stool sample will also be collected 2-3 months after the first for a sub-sample of N=300 to assess intra-individual variability in microbiota profiles. The selected participants will receive a stool self-sampling kit with detailed instructions by post to their home address. The pseudonymized samples will be returned by mail by the participant to the processing laboratory, which will determine their gut microbiota characteristics by 16S rDNA sequencing and/or " shotgun " sequencing. The gut microbiota profiles will then be analyzed in a pseudonymised manner in association with diet and health, using data collected as part of the NutriNet-Santé cohort follow-up (e.g. food consumption, prevalence and incidence of pathologies, biological data, anthropometric characteristics, medication intake, socio-demographic characteristics, lifestyle).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the NutriNet-Santé cohort
* Age ≥ 18 years
* Resident of metropolitan France
* Written comprehension frenc

Exclusion Criteria:

* Person subject to a safeguard of justice measure
* Person belonging to one of the categories of vulnerable persons
* Diagnosis of COVID-19 (clinically or by PCR) in the month prior to collection
* Contact with a COVID-19 patient in the month prior to collection
* Suspicion of COVID-19 in the month preceding collection (clinical signs of infection : fever associated with headache, respiratory signs, os anosmia/ageusia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2033-12-15 (Estimated); Study Completion 2033-12-15 (Estimated)

PRIMARY OUTCOMES:
Characterization of gut microbiota profile by 16S r RNA gene sequencing | At inclusion, 2 to 3 months later
  Performed on self sampling of stools at home. It is used to characterize the taxonomic profiles of intestinal microbiota. It will be applied on all samples
Characterization of gut microbiota profile by " shotgun " metagenomic sequencing | At inclusion, 2 to 3 months later
  Performed on self sampling of stools at home. It provides more detailled characterization of the taxonomic and functional profiles of the intestinal microbiota. It will be applied to a smaller number of samples (no more than 300).

CONTACTS AND LOCATIONS:
Locations (1):
- EREN SMBH Université Sorbonne Paris Nord, Bobigny, France

IPD SHARING:
Plan to Share IPD: No